CLINICAL TRIAL: NCT00804349
Title: Apnea Rampant In Acute Decompensated Heart Failure II
Brief Title: Treatment of Sleep Disordered Breathing In Acute Decompensated Heart Failure Patients
Acronym: ARIA-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Nexan Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HN-3025
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2013-02

CONDITIONS: Heart Failure; Sleep Apnea Syndromes
Keywords: Heart Decompensation; Heart Failure, Congestive; Heart Failure, Left-Sided; Heart Failure, Right-Sided; Apnea, Sleep; Sleep Apnea, Mixed Central and Obstructive; Sleep Hypopnea; Sleep-Disordered Breathing
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients will receive standard medical therapy for heart failure only and will not receive Autotitrating Positive Airway Pressure therapy.
- Autotitrating Positive Airway Pressure (Active Comparator): Patients will receive Autotitrating Positive Airway Pressure therapy in addition to standard medical care for heart failure.
  Interventions: Device: Autotitrating Positive Airway Pressure

INTERVENTIONS:
Device: Autotitrating Positive Airway Pressure — Patients will be treated with Autotitrating Positive Airway Pressure therapy
  Arms: Autotitrating Positive Airway Pressure

SUMMARY:
Heart Failure affects 5-6 million Americans and there are about 550 thousand new cases of heart failure every year. There are approximately 3 million hospital admission for acute decompensated heart failure with hospital readmission rate of 20% at 30 days and 50% at 60 day, costing up to 20 billion dollars per year. In our previous study we have discovered that sleep disordered breathing is prevalent in 70% of patients with acute decompensated heart failure. We hypothesize that, detection and treatment of sleep disordered breathing in acute decompensated heart failure patients will reduce episodic hypoxic events during acute decompensation and may decrease hospital length of stay and reduce future readmissions.

DETAILED DESCRIPTION:
Background:

Heart failure (HF) affects 5 to 6 million Americans and is increasing in prevalence. There are about 550,000 new cases of heart failure every year and about 3 million admissions for acute decompensated heart failure every year. Despite advances in medical care, the hospital readmission rate is 20% at one month and 50% at six months. The total cost of heart failure on the health system is upwards of 35 billion dollars per year. About half of these resources are used during acute hospitalizations.

An important limitation to the current approach to the management of HF is the focus on the awake patient. This approach underestimates the mechanisms that might contribute to the pathophysiology or progression of HF.

Sleep disordered breathing (SDB) is very common in congestive heart failure. Recently, the adverse implications of SDB in patients with HF have been appreciated. Intermittent apnea-induced hypoxia, hypercapnia, surges in central sympathetic outflow and left ventricular afterload, daytime hypertension, and loss of vagal heart rate regulation are potent stimuli to myocyte necrosis and apoptosis, myocardial ischemia, arrhythmias, adverse cardiac remodeling, and the resulting accelerated disease progression in HF.

This makes us believe that treatment of SDB during acute decompensated heart failure in addition to standard medical therapy (SMT) would be beneficial.

Study Design:

80 eligible patients admitted to Albert Einstein Medical Center with the diagnosis of Acutely Decompensated Heart Failure will be recruited for the study. Once patients have been identified, inclusion and exclusion criteria met, they will be consented to participate in the trial within 24 to 48 hours of admission to the hospital. After enrollment, the patient will be screened for SDB with NEXAN CPS system. The Sensor, a flexible data collection patch that adheres to the patient's chest, continuously records ECG, respiratory, and oximetry data and allows for future use and evaluation. Patients with SDB will be further randomized to SDB monitoring only and SDB monitoring plus Autotitratable Continuous Positive Airway Pressure (APAP) treatment arm. Patients in both arms will be treated with standard of care therapy for acute heart failure. There is a possibility that patients randomized to APAP therapy may refuse further treatment after the first night. These patients will be analyzed on the basis of intention to treat approach

Once randomized, all patients will be fitted with the NEXAN Clear Path System and will continue to wear it until the time of discharge or 7 days. Those in the treatment group will be fitted with an Autotitratable Continuous Positive Airway Pressure device and will be continued on treatment until discharged or a maximum of 7 days.

Follow-up of these patients will include a 15 day and 60 day phone call and a 30 day office visit. At the 30 day visit the patients will be asked to use the NEXAN sensor for that night, and return the equipment the next day. The patients that were determined to have sleep-disordered breathing will be referred for a full overnight polysomnography test.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 and able to consent
* NYHA Class III/IV Symptoms
* Objective Evidence of Heart Failure
* Physical Exam consistent with Heart Failure
* BNP greater than 500
* Radiographic Evidence of Heart Failure
* SDB (AHI > 5/hour) on Nexan CPS
* Ability to tolerate appropriate medical therapy for Heart Failure
* Willingness to follow-up as an outpatient after discharge

Exclusion Criteria:

* Patients with known Sleep-Disordered Breathing currently using CPAP or BiPAP
* Patients with known COPD
* Patients with known restrictive lung disease
* Patients with tracheostomy in place
* Acute MI/Acute Coronary Syndrome at time of hospitalization
* Cardiogenic Shock
* Troponin Leak greater than 0.08
* Patients with major multisystem disorders
* Expected survival less than 6 months
* End Stage Renal Disease on Dialysis
* Chronic Liver Disease
* Albumin level less than 3.
* Patients from Nursing homes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darshak Karia, MD, Principal Investigator — Albert Einstein Medical Center. Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.
Pre-assignment Details: 0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.
Groups:
- Control: Patients will receive standard medical therapy for heart failure only and will not receive Autotitrating Positive Airway Pressure therapy.
  0 participants analyzed. The study was closed and the PI is not longer at the institution. The PI was contacted to complete requirements but the information was not added by the PI. No study data are available.
- Autotitrating Positive Airway Pressure: Patients will receive Autotitrating Positive Airway Pressure therapy in addition to standard medical care for heart failure.
  Autotitrating Positive Airway Pressure: Patients will be treated with Autotitrating Positive Airway Pressure therapy
  0 participants analyzed. The study was closed and the PI is not longer at the institution. The PI was contacted to complete requirements but the information was not added by the PI. No study data are available.
Period: Overall Study
Arm/Group | Control | Autotitrating Positive Airway Pressure
Started | 0 (0 analyzed PI no longer at institution;PI contacted, information not added; No data available.) | 0 (0 analyzed PI no longer at institution;PI contacted, information not added; No data available)
Completed | 0 (0 analyzed PI no longer at institution;PI contacted, information not added; No data available) | 0 (0 analyzed PI no longer at institution;PI contacted, information not added; No data available)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.
Groups:
- Control: Patients will receive standard medical therapy for heart failure only and will not receive Autotitrating Positive Airway Pressure therapy.
  0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.
- Autotitrating Positive Airway Pressure: Patients will receive Autotitrating Positive Airway Pressure therapy in addition to standard medical care for heart failure.
  Autotitrating Positive Airway Pressure: Patients will be treated with Autotitrating Positive Airway Pressure therapy
  0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.
- Total: Total of all reporting groups
Arm/Group | Control | Autotitrating Positive Airway Pressure | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Episodic Oxygen Desaturation
Description: 0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.
Time Frame: Concurrent
Population: as for baseline characteristics
Arm/Group | Control | Autotitrating Positive Airway Pressure
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Readmission
Description: as for outcome 1
Time Frame: 30 days post discharge
Population: as for baseline characteristics
Arm/Group | Control | Autotitrating Positive Airway Pressure
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Length of Stay
Description: as for outcome 1
Time Frame: Concurrent
Population: as for baseline characteristics
Arm/Group | Control | Autotitrating Positive Airway Pressure
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Visual Analog Scale of Shortness of Breath
Description: as for outcome 1
Time Frame: Concurrent
Population: as for baseline characteristics
Arm/Group | Control | Autotitrating Positive Airway Pressure
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.
Description: 0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.
Arm/Group | Control | Autotitrating Positive Airway Pressure
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
0 participants analyzed. Study closed; PI no longer at the institution. Efforts to have the PI add the required information have been unsuccessful. No study data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No